CLINICAL TRIAL: NCT01115907
Title: Clinical Investigation of the Freedom SOLO Stentless Heart Valve in North America
Brief Title: Freedom SOLO Stentless Heart Valve Study
Acronym: SOLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G100014
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Aortic Stenosis; Aortic Insufficiency
Keywords: Aortic; Valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Freedom SOLO stentless valve implant (Experimental): Appropriate subjects will receive the Freedom SOLO stentless valve implant as a replacement for a diseased or damaged native or prosthetic aortic valve.
  Interventions: Device: Freedom SOLO Stentless Heart Valve

INTERVENTIONS:
Device: Freedom SOLO Stentless Heart Valve — Freedom SOLO Stentless Heart Valve

SUMMARY:
The purpose of this clinical investigation is to demonstrate the safety and effectiveness of the Freedom SOLO heart valve.

DETAILED DESCRIPTION:
The SOLO clinical investigation is a prospective, non-randomized, multicenter trial of the SOLO Freedom heart valve implanted in patients requiring aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female 18 years old or older.
* The subject or subject's legal representative is willing to sign the informed consent.
* The subject which preoperative evaluation indicated the need for native or prosthetic aortic valve replacement.
* Any subject amenable to aortic valve replacement with biological prosthesis should be enrolled in the study, even in conjunction with valve repair, coronary artery bypass grafting and other procedures.
* The subject is located in a geographic location that will enable the subject to return to the study site for all follow-up examinations (i.e. geographically stable).
* Subject will be available to the investigator(s) for postoperative follow-up beyond one year.

Exclusion Criteria:

* The subject has preexisting valve prosthesis in the mitral, pulmonary or tricuspid position.
* The subject requires a double or multiple valve replacement (a valve repair is not considered an exclusion criterion).
* The subject has a previously implanted SOLO valve, within the clinical study, that requires replacement.
* The subject has active endocarditis or myocarditis.
* The subject is or will be participating in a concomitant research study of an investigational product.
* The subject is a minor, drug abuser, alcohol abuser, prison inmate, institutionalized, or is unable to give informed consent.
* The subject has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy of less than 1 year, or the implant of the device produces an unacceptable increased risk to the subject.
* The subject is pregnant, planning to become pregnant or lactating.
* The subject has a congenital bicuspid aortic valve.
* The subject is known to be noncompliant or is unlikely to complete the study.
* The subject is undergoing renal dialysis for chronic renal failure or has been diagnosed with hyperparathyroidism.
* The subject has had an acute preoperative neurological deficit, myocardial infarction, or cardiac event that has not returned to baseline or stabilized ≥30 days prior to the planned valve implant surgery.
* The subject has extensive calcification of the aortic root where removal of the calcified tissue cannot be achieved.
* The subject has a significantly dilated aortic root that is not surgically corrected.
* The subject requires replacement of the aortic root / full root procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety will be determined by incidence rate of adverse events | 1 year
  The complication and survival rates for the SOLO valve are comparable to appropriate historical controls manifested as objective performance criteria (OPCs) and to that reported in the literature for other stentless bioprostheses and stented pericardial valves.

SECONDARY OUTCOMES:
Efficacy will be determined by hemodynamics | 1 year
  The hemodynamic performance of the SOLO valve will be compared to that reported in the literature for other stentless bioprostheses and stented pericardial valves.
Effectiveness will be determined by NYHA Classification comparisons | 1 year
  Clinically significant improvement in overall patient condition by comparison of preoperative and postoperative NYHA functional classifications.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, M.D., Principal Investigator — The Cleveland Clinic; David Heimansohn, MD, Principal Investigator — St. Vincent Heart Center; Alex Zapolanski, MD, Principal Investigator — The Valley Hospital; Vinod Thourani, MD, Principal Investigator — Emory University; Reza Dabir, MD, Principal Investigator — Oakwood Hospital; Ali Khoynezhad, MD, Principal Investigator — Cedars-Sinai Medical Center; Pranshanth Vallabhajosyula, MD, Principal Investigator — University of Pennsylvania; Michael Moront, MD, Principal Investigator — The Toledo Hospital; Scott Goldman, MD, Principal Investigator — Main Line Health; Shaohua Wang, MD, Principal Investigator — University of Alberta; L. Ray Guo, MD, Principal Investigator — London Health Science Centre; Andrew Maitland, MD, Principal Investigator — Foothills Medical Center; Michael Moon, MD, Principal Investigator — St. Boniface Hospital; Pierre Voisine, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval; Jian Ye, MD, Principal Investigator — St. Paul's Hospital
Locations (15):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Oakwood Hospital, Dearborn, Michigan
  - The Valley Hospital, Ridgewood, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Bristish Columbia St. Paul Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec